CLINICAL TRIAL: NCT05717114
Title: Efficacy of Different Doses of Dexmetomedine as an Adjuvant to Bupivacaine in Ultrasound Guided PECS Block in Patients Undergoing Modified Radical Mastectomy
Brief Title: Dexmetomedine as an Adjuvant to Bupivacaine in Ultrasound Guided PECS Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, rabab Mohammad habeeb, Principal investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1/2023,ANET2-1
Record Dates: First submitted 2023-01-23; First posted 2023-02-08 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Prospective randomized study
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Placebo Comparator): received plan bupivacaine1ml/Kg
  Interventions: Procedure: Pecs block
- Group II (Active Comparator): received plain bupivacaine 1ml/Kg plus dexmetomedine0.5 µg/Kg
  Interventions: Procedure: Pecs block
- GroupIII (Active Comparator): received plain bupivacaine 1ml/Kg plus dexmetomedine1µg/Kg
  Interventions: Procedure: Pecs block

INTERVENTIONS:
Procedure: Pecs block — (Pecs block):the block will be performed with the patients in the supine position.The infraclavicular and axillary regions will be cleaned with antiseptic solution. the inplane technique will be used from proximal and medial to distal and lateral in an oblique manner at dermatome level T2and T3.The puncture site was infiltrated with 2%lidocaine and once the structures is identified with ultrasound.

SUMMARY:
Regional anesthesia is an essential component of anesthesia and analgesia. It has many advantages, it decreases pain post operatively, improves patient outcome and allow early recovery and ambulation Post-operative pain following breast surgery results from injured muscles and nerves, management of acute post operative pain is a consistent factor for better outcome and patient satisfaction

DETAILED DESCRIPTION:
All patients will be monitored by standard intraoperative monitoring that includes continuous electrocardiography (ECG), capnography, pulse oximetry, and non invasive blood pressure.

Induction of general anesthesia will be done by propofol 1.5-2 mg/kg and fentanyl 3µg/kg.

Tracheal intubation will be facilitated by administration of rocuronium 0.8 mg/kg. Anesthesia will be maintained with isoflurane 1MAC (Pecs block):the block will be performed with the patients in the supine position.The infraclavicular and axillary regions will be cleaned with antiseptic solution. the in plane technique will be used from proximal and medial to distal and lateral in an oblique manner at dermatome level T2 and T3.The puncture site was infiltrated with 2%lidocaine and once the structures is identified with Ultrasound

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* aged 18-60years old
* ASA class 1 to 3
* scheduled for elective modified radical mastectomy

Exclusion Criteria:

* patients refusal,
* coagulopathies
* concurrent anticoagulant therapy
* allergy to local anaesthetics
* infection at puncture site

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females understanding Mastectomy
Enrollment: 96 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 48 hours
  Visual analog score for pain where 0 no pain and 10 most severe pain

SECONDARY OUTCOMES:
Total morphine consumption | 48 hours
  Mg

CONTACTS AND LOCATIONS:
Overall Officials: rabab M habeeb, Principal Investigator — Menoufia University
Locations (1):
- Menoufia, Menoufia, Monufia Governorate, Egypt